CLINICAL TRIAL: NCT02452255
Title: Mechanisms of Fenofibrate and Propranolol Alone or Combined in Burn Patients
Brief Title: Fenofibrate and Propranolol in Burn Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Shriner's Burn Hospital closed the study and access to study-related data is unavailable. We are unable to submit the additional information or results-data
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Shriners Hospitals for Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-0441; NIH RO1GM056687 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2015-05-12; First posted 2015-05-22 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2018-08

CONDITIONS: Burn
MeSH Terms: conditions — Burns | interventions — Fenofibrate; Propranolol; Metoprolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fenofibrate (Active Comparator): Fenofibrate by mouth given daily throughout hospitalization for up to 12 months
  Interventions: Drug: Fenofibrate
- Fenofibrate and Propranolol (Active Comparator): Fenofibrate and Propranolol by mouth given throughout hospitalization for up to 12 months
  Interventions: Drug: Fenofibrate; Drug: Propranolol
- Placebo (Placebo Comparator): Placebo by mouth given daily throughout hospitalization for up to 12 months.
  Interventions: Drug: Placebo
- Propranolol (Active Comparator): Propranolol by mouth given throughout hospitalization for up to 12 months
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Fenofibrate — Fenofibrate by mouth given daily throughout hospitalization for up to 12 months
  Other Names: Tricor
  Arms: Fenofibrate; Fenofibrate and Propranolol
Drug: Placebo — Placebo by mouth given daily throughout hospitalization for up to 12 months
  Other Names: Control
  Arms: Placebo
Drug: Propranolol — Propranolol by mouth given daily throughout hospitalization for up to 12 months
  Other Names: Metoprolol; inderal
  Arms: Fenofibrate and Propranolol; Propranolol

SUMMARY:
The proposed study will test the hypothesis that Propranolol, fenofibrate and fenofibrate plus propranolol have therapeutic, physiological, and metabolic effects that will improve clinical outcomes, and the long-term recovery, rehabilitation, and QOL in burned patients.

DETAILED DESCRIPTION:
Determine the clinical benefits and underlying mechanisms whereby the metabolic perturbators fenofibrate and propranolol impact burn patient outcomes. The investigators hypothesize that these metabolic regulators given for one year will maintain body mass, improve muscle function by increasing protein synthesis, augment wound healing, reduce fibrosis, improve cardiovascular function, reduce systemic inflammation, restore insulin sensitivity, and decrease liver dysfunction without the risk of the hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* 0 through 80 years
* ≥ 20% Total Body Surface Area Burn injury

Exclusion Criteria:

Pregnancy

History or existence of pre-burn injury conditions

* Allergies to propranolol or fenofibrate
* Asthma requiring treatment
* Congestive heart failure (measured ejection fraction < 20%)
* Renal or hepatic disease
* Medical condition requiring glucocorticoid treatment
* History of AIDS, Aids Related Complex or HIV
* History of Cancer within 5 years

Decision not to treat due to burn injury severity or futility as deemed by the clinical team

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Glucose Metabolism | From randomization up to one year
  Glucose levels and amount of regular insulin infused during hospitalization.

SECONDARY OUTCOMES:
Hypermetabolism | From randomization up to one year
  Resting energy expenditure (REE) done weekly while in hospital
Rate pressure product | Participants will be followed for the duration of hospital stay, an average of 5 weeks
  Multiply the subjects resting heart rate and systolic blood pressure measurements and average every 24 hours while hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — University of Texas
Locations (1):
- Shriners Hospitals for Children, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No